CLINICAL TRIAL: NCT07266649
Title: Effects of Pilates Training on Ankle Proprioception, Postural Control and Performance in Footballers With Chronic Ankle Instability
Acronym: CAI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/020
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Proprioception, Postural Balance; Performance; Chronic Ankle Instability, CAI
Keywords: Chronic Ankle Instability; proprioception; Postural Control; Performance
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, the blinding of participants and therapist was not feasible. To overcome the assessment bias, the outcome assessor remained blinded to group allocations, maintain single blinded study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Pilates training group
  Interventions: Other: Pilates exercises
- Group B (Experimental): Balance training group
  Interventions: Other: Balance exercises

INTERVENTIONS:
Other: Pilates exercises — Duration: 8 weeks (3 sessions/week) Session Duration: 60 minutes per session Equipment Used: Yoga mat, resistance bands, Pilates ring, small stability ball, foam roller.
  Structure of Each Session:
  Phase Time Activities Warm-Up 10 min Gentle dynamic stretches and mobility exercises (e.g., neck rolls, shoulder circles, hip openers, ankle circles) Core Pilates Training 40 min - Beginner-Intermediate Mat Pilates targeting core, hips, gluts, and lower leg muscles - Sample Exercises: - Pelvic tilts - Hundred - Single-leg stretch - Shoulder bridge with ankle engagement - Side-lying leg circles - Toe taps and leg lifts with ankle focus Cool Down 10 min Static stretching, deep breathing, and relaxation techniques
  Progression:
  Exercises will be progressed weekly by:
  * Increasing repetitions and sets
  * Reducing support (e.g., double leg to single leg)
  * Incorporating dynamic and unstable surfaces (foam pads, balance discs)
  Arms: Group A
Other: Balance exercises — Group B: Control Group Duration: 8 weeks (3 sessions/week) Session Duration: 60 minutes per session Equipment Used: Balance board, wobble disc, cones, foam pads, resistance bands.
  Structure of Each Session:
  Phase Time Activities Warm-Up 10 min Light jogging, ankle mobility drills, dynamic stretching Balance Training 40 min - Static and Dynamic Balance Drills: - Single-leg stance (eyes open/closed) - Wobble board balancing - Star excursion balance test practice - Tandem walking on a line - Forward/backward hops on one leg - Cone drills with reach tasks and steps up Cool Down 10 min Ankle and lower limb stretching, breathing techniques
  Progression:
  * Decrease base of support
  * Introduce perturbations (e.g., partner tapping)
  * Dual-task activities (catching, counting, etc.)
  Arms: Group B

SUMMARY:
This study aims to contribute to the effects of Pilates training on ankle proprioception, postural control, and performance in football players with chronic ankle instability. Eighty eight participants will be randomly allocated into two groups and will receive both Pilates and balance training for eight weeks. it is hypothesized that the group that will receive Pilates taring will produce greater improvements as compared to other group.

DETAILED DESCRIPTION:
Chronic ankle instability is a frequently encountered issue in footballers, characterized by repeated episodes of the ankle "giving way," resulting in functional limitations and increased risk of future injuries. Conventional rehabilitation protocols often fail to restore optimal neuromuscular control, particularly proprioceptive and postural capabilities. Given the demands of football, this deficit can significantly hinder athletic performance and increase injury susceptibility. While Pilates-based rehabilitation has shown promise in improving core strength, balance, and neuromuscular coordination, there is a paucity of research examining its role in the context of CAI. This study addresses this research gap by assessing the effectiveness of Pilates training in improving key functional deficits among footballers with CAI, potentially informing more effective and sport-specific rehabilitation strategies.

Participants will be randomized into two groups:

1. Pilates Training Group
2. Control Group Intervention The intervention will last [insert duration 8 weeks], with participants attending three supervised sessions per week. Each session will last 60 minutes and will be led by a qualified physical therapist experienced in Pilates and sports rehabilitation.

After the intervention period, post-intervention assessments using the same outcome tools will be conducted by the same blinded assessor under identical conditions to the baseline evaluation. Any adverse events or dropouts will be recorded throughout the study.

Group A: Pilates Intervention Group Duration: 8 weeks (3 sessions/week) Session Duration: 60 minutes per session Equipment Used: Yoga mat, resistance bands, Pilates ring, small stability ball, foam roller.

Structure of Each Session:

Phase Time Activities Warm-Up 10 min Gentle dynamic stretches and mobility exercises (e.g., neck rolls, shoulder circles, hip openers, ankle circles) Core Pilates Training 40 min - Beginner-Intermediate Mat Pilates targeting core, hips, gluts, and lower leg muscles - Sample Exercises: - Pelvic tilts - Hundred - Single-leg stretch - Shoulder bridge with ankle engagement - Side-lying leg circles - Toe taps and leg lifts with ankle focus Cool Down 10 min Static stretching, deep breathing, and relaxation techniques

Progression:

Exercises will be progressed weekly by:

* Increasing repetitions and sets
* Reducing support (e.g., double leg to single leg)
* Incorporating dynamic and unstable surfaces (foam pads, balance discs) Group B: Control Group Duration: 8 weeks (3 sessions/week) Session Duration: 60 minutes per session Equipment Used: Balance board, wobble disc, cones, foam pads, resistance bands.

Structure of Each Session:

Phase Time Activities Warm-Up 10 min Light jogging, ankle mobility drills, dynamic stretching Balance Training 40 min - Static and Dynamic Balance Drills: - Single-leg stance (eyes open/closed) - Wobble board balancing - Star excursion balance test practice - Tandem walking on a line - Forward/backward hops on one leg - Cone drills with reach tasks and steps up Cool Down 10 min Ankle and lower limb stretching, breathing techniques

Progression:

* Decrease base of support
* Introduce perturbations (e.g., partner tapping)
* Dual-task activities (catching, counting, etc.)

ELIGIBILITY:
Inclusion Criteria:

Male footballers aged 22-35

* History of unilateral ankle sprain in past 12 months
* Inability to bear weight post-injury
* CAIT score < 24
* Minimum of 1-year experience in football

Exclusion Criteria:

* Bilateral ankle sprains
* Lower limb fractures or surgeries
* Neurological conditions (e.g., MS, CMT, Stroke)

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 88 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Postural control | Base line before intervention after 8 weeks post intervention
  The YBT has the patient stand on one leg while reaching out in 3 different directions with the other lower extremity. They are anterior, posteromedial and posterolateral. When using the Y-Balance test kit, the 3 reaches yield a "composite reach distance" or composite score used to predict injury.
ankle proprioception | Baseline: Before intervention 8 weeks post-intervention
  The goniometer was used to measure the ankle proprioception. Testing was performed the way that the person would sit on a chair so that a 90-degree angle of thigh and knee was maintained, and the height of the chair was such that the soles of the individual could not reach the ground. Then the person's foot was positioned with the goniometer in such a way that the eyes of the person were closed. Then the individual foot was inactively taken to the midrange. This angle was 10 degrees for dorsiflexion, 20 degrees for plantar flexion, 15 degrees for inversion and 10 degrees for eversion. Afterwards, the person was asked to actively re-create the desired angle with his closed eye; the test was performed three times, and the mean of three times of the angle of reconstruction determined the individual's score in each of the state.
performance | base line before intervention and 8 weeks post intervention
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. This self-report outcome instrument is available in English, German, French and Persian. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: The Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale. The Sports subscale assesses more difficult tasks that are essential to sport, it is a population-specific subscale designed for athletes.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tariq Shafi, Study Chair — Lahore University of Biological and Applied Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghorbani M, Yaali R, Sadeghi H, Granacher U. Effects of Pilates Exercise Training on Static Balance and Lower Limbs Proprioception in Adult Females With and Without Flexible Flatfeet. Foot Ankle Spec. 2024 Sep 26:19386400241279930. doi: 10.1177/19386400241279930. Online ahead of print. PMID 39324770
- [Background] Zhang C, Chen N, Wang J, Zhang Z, Jiang C, Chen Z, Fang J, Peng J, Li W, Song B. The Prevalence and Characteristics of Chronic Ankle Instability in Elite Athletes of Different Sports: A Cross-Sectional Study. J Clin Med. 2022 Dec 16;11(24):7478. doi: 10.3390/jcm11247478. PMID 36556094
- [Background] Alghadir AH, Iqbal ZA, Iqbal A, Ahmed H, Ramteke SU. Effect of Chronic Ankle Sprain on Pain, Range of Motion, Proprioception, and Balance among Athletes. Int J Environ Res Public Health. 2020 Jul 23;17(15):5318. doi: 10.3390/ijerph17155318. PMID 32718066
- [Background] Ziaei Ziabari E, Haghpanahi M, Razi M, Lubberts B, Ashkani-Esfahani S, DiGiovanni CW. The Effects of Chronic Ankle Instability on the Biomechanics of the Uninjured, Contralateral Ankle During Gait. Orthop Surg. 2022 Sep;14(9):2238-2244. doi: 10.1111/os.13307. Epub 2022 Jul 19. PMID 35852096
- See also: Related Info — https://www.researchgate.net/publication/387477246_EFFECTS_OF_PILATES_EXERCISES_ON_BALANCE_AND_GAIT_IN_SCHOOL_GOING_CHILDREN